CLINICAL TRIAL: NCT02670226
Title: Metabolomics and Transcriptomics Approaches to Identify Muscular Biomarkers in Amyotrophic Lateral Sclerosis
Brief Title: Muscular Biomarkers in Amyotrophic Lateral Sclerosis
Acronym: METABOMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO15-HB-METABOMU; 2015-A01629-40 (Other: IdRCB); 151550B-31 (Other: ASNM); 2016-R3 (Other: CPP)
Record Dates: First submitted 2016-01-14; First posted 2016-02-01 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Muscle metabolism; Metabolomics; Transcriptomics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case group (Other): The intervention, specific to the study, is to take samples at baseline on patients with Amyotrophic Lateral Sclerosis
  Interventions: Other: Samples
- Control group (Other): The intervention, specific to the study, is to take samples at baseline on patients without neurological disease
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood samples, muscle biopsy

SUMMARY:
The first objective is to find some biomarkers, or a profile of biomarkers of ALS to help to diagnosis. The second objective is to better understand the pathogenesis of this disease by the exploration of muscle, blood and satellite cells metabolomes and transcriptomes.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS), the most common MND, is a fatal adult-onset neuromuscular disease. Due to clinical heterogeneity and absence of biological tools to diagnose ALS, the delay between the first symptoms and diagnosis averages 9-13 months. A group of pathophysiological processes, including oxidative stress and glutamate-mediated excitotoxicity contribute to cell death, but the triggering factor, the timing and the interaction of different cellular events await elucidation [2]. Unknown pathogenesis for most patients means few available treatments. The search for biomarkers that can aid diagnosis, characterize phenotype, define pathophysiology, identify endpoints in trials and measure disease progression is of utmost importance for the field. Some studies have advocated that muscle per se may be impaired by pathogenesis of the diseases. Muscle has been poorly studied and its central role in energetic metabolism suggests that this tissue, quite easily available, should be more analyzed to find biomarkers and to compare muscular metabolism with those of brain and overall body. Specific aims of our subjects are:

Specific aims are focused on:

1. the acquisition of metabolites profiles of the muscle, blood and satellite cells using an analytical platform enable a deep exploration. For that, the use of three analytical modalities (NMR, mass spectrometry coupled to GC or UPLC) ensures the best coverage of the metabolite population with a high range of concentration variability and molecular diversity.
2. the building of metabolites profiles models that discriminate pathological and control situations.
3. the identification of metabolites implicated in the discriminant model.
4. the generation of metabolism pathways hypothesis related to the discriminant model.
5. the acquisition of transcriptomics data to confirm and add complementary results to metabolomics data

ELIGIBILITY:
Case group selection criteria:

Inclusion Criteria:

* Age ≥ 18 years and ≥ 75 years
* ALS according to the El Escorial criteria
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindication to biopsy
* Contraindication to local anesthesia
* Treatment with oral or injectable anticoagulants, antiplatelet (except aspirin)
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Treatment against cramps or twitching may affect muscle metabolism

Control group selection criteria:

Inclusion Criteria:

* Age ≥ 18 years and ≥ 75 years
* No neuronal disease
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindication to biopsy
* Treatment with oral or injectable anticoagulants, antiplatelet (except aspirin)
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Treatment against cramps or twitching may affect muscle metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Metabolic signature of muscle | At baseline
  Metabolomics profile using NMR and LC-HRMS
Metabolic signature of blood | At baseline
  Metabolomics profile using NMR and LC-HRMS
Metabolic signature of satellites cells | At baseline
  Metabolomics profile using NMR and LC-HRMS

SECONDARY OUTCOMES:
Expression levels of targeted genes using transcriptomics | At baseline
  Choice of genes based on results obtained by metabolomics approaches

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BLASCO, MD, Study Director — helene.blasco@univ-tours.fr
Locations (2):
- France (2):
  - Service de chirurgie orthopédique et traumatologique, CHRU de TOURS, Tours
  - Service de Neurologie, CHRU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lanznaster D, Bruno C, Bourgeais J, Emond P, Zemmoura I, Lefevre A, Reynier P, Eymieux S, Blanchard E, Vourc'h P, Andres CR, Bakkouche SE, Herault O, Favard L, Corcia P, Blasco H. Metabolic Profile and Pathological Alterations in the Muscle of Patients with Early-Stage Amyotrophic Lateral Sclerosis. Biomedicines. 2022 Jun 2;10(6):1307. doi: 10.3390/biomedicines10061307. PMID 35740329